CLINICAL TRIAL: NCT05877040
Title: Anti-nerve Reactivity as Predictor of Response to Immune Therapy in Patients With Chronic Inflammatory Demyelinating Polyradiculoneuropathy (CIDP): A Proof of Concept Study With Rituximab in Patients With CIDP Not Responding to Conventional Immune Therapy
Brief Title: A Proof of Concept Study With Rituximab in Patients With CIDP Not Responding to Conventional Immune Therapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RF-2016-02361887
Record Dates: First submitted 2023-05-17; First posted 2023-05-26 (Actual); Last update posted 2023-05-26 (Actual); Status verified 2023-05

CONDITIONS: Polyradiculoneuropathy, Chronic Inflammatory Demyelinating
MeSH Terms: conditions — Polyradiculoneuropathy, Chronic Inflammatory Demyelinating | interventions — Rituximab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treated (Experimental)
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Rituximab — Open label proof-of-concept study with intravenous Rituximab, given at the dose of 1g in one day, followed by the same dose after two weeks

SUMMARY:
Chronic inflammatory demyelinating polyradiculoneuropathy (CIDP) is a chronic and often disabling neuropathy that often responds to immune therapies. A few phenotypes have been identified even if it is unclear whether they are variants of CIDP or different diseases considering their relatively different responses to therapy. Antibodies against proteins at the node of Ranvier, including contactin 1 and neurofascin 155, have been reported in up to 10% of the patients and were associated to a poor response to CIDP therapy but a positive response to Rituximab supporting the heterogeneity of CIDP. We will examine these antibodies in a large population of Italian CIDP patients included in a Database and correlate their presence with the clinical and electrophysiological features of the neuropathy, its progression and response to therapy. We will perform an open label prospective therapeutic study with Rituximab in patients with CIDP not responsive to conventional immune therapies and will correlate the response to therapy to the clinical phenotype and the presence of anti-neural antibodies.This may lead to a more appropriate choice of therapy in CIDP avoiding the use of expensive and possibly ineffective therapy. We will also collect the biological samples (serum and when available CSF) of the patients with CIDP and store them to allow the formation of a biological bank that may be used in future immunological studies to clarify the pathogenesis a of the disease and possibly to identify biomarkers of the disease and of response to therapy. This study will permit to collect a sufficiently large number of adequately and homogeneously examined patients with CIDP, with different antibody reactivities and with unsatisfactory response to therapy. This will permit to have sufficiently large number of patients to perform an open-label study with Rituximab whose efficacy has been so far reported only in anecdotal reports on small number of patients.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is ≥ 18 years of age at Visit1 (screening) and who signed the informed consent form for the study
2. Subject has a documented diagnosis of definite or probable CIDP according to the EFNS/PNS criteria 2010 (Joint Task Force of the EFNS and the PNS, 2010)
3. Subject has not improved after and adequate dose of therapy with intravenous immunoglobulins (IVIg) corresponding to at least 2 g/kg monthly for two months, steroids corresponding to the equivalent of at least 1 mg/kg daily of oral prednisone for two months or a course of at least 4 plasma exchanges within two weeks.
4. Subject can take steroids at the maximum dosage equivalent to 25 mg/day of prednisone or pulsed 600 mg/monthly of methylprednisolone as far as the dosage has not been increased (+ 20%) in the previous 6 months and has not determined a satisfactory response to therapy.
5. Female subjects of childbearing potential according with the CTFG guidelinesa must have a negative serum pregnancy test and agree to use a highly effective method of birth control in accordance with the CTFG guidelinesb during the study and for a period of 12 months after their last dose of study drug.
6. Male subject, when sexually active, with a partner of childbearing potential according with the CTFG guidelinesa must be willing to use a highly effective method of birth control in accordance with the CTFG recommendationsb during the study and for 12 months after the final administration of rituximab.

Exclusion Criteria:

Subject has a current diagnosis or has a history of Type 1 or Type 2 diabetes mellitus 2. Subject has IgM paraproteinemia with anti-myelin associated glycoprotein antibodies 3. Subject has Multifocal Motor Neuropathy with conduction block (MMN) 4. Clinical or known evidence of associated medical conditions that might cause neuropathy, including but not limited to connective tissue disease, Lyme disease, cancer (with the exclusion of benign skin cancer), Castleman's disease and systemic lupus erythematosus, malignant plasma cell dyscrasia, lymphoma, osteosclerotic myeloma, POEMS, or assumption of agents that may lead to neuropathy (eg, amiodarone therapy).

5. Female who is pregnant or lactating 6. Subjects with any medical or psychiatric condition (acute or chronic) that, in the opinion of the investigator, could harm the subject or would compromise the subject's ability to participate in the study.

7. Subjects with congestive heart failure or a moderate or severe impairment of cardiac function 8. Subjects with renal impairment defined as: serum creatinine > 1.4 mg/dL for females and 1.5 mg/dL for males 9. Subjects with an absolute leukocyte count <4000/mm3, lymphocyte count <800/mm3, platelet count <100,000/mm3 10. Subjects with liver impairment defined as total or conjugated bilirubin >1.5 × upper limit of the normal (ULN) range, unless in context of Gilbert's syndrome; aspartate aminotransferase (AST), alanine aminotransferase (ALT) >3 × ULN range; alkaline phosphatase (AP) >1.5 × ULN range; gamma-glutamyl-transferase (GGT) >3 × ULN range 11. Subjects with a history of clinically relevant ongoing chronic infections including but not limited to human immunodeficiency virus (HIV), hepatitis B, hepatitis C, active or latent tuberculosis or is tested positive for HIV (anti-HIV1 or anti-HIV2 antibodies) hepatitis B (HBsAG positive or HBcAb positive without HBsAb) or hepatitis C (HCV antibodies) at the screening visit.

12. Subject has a family history of primary immunodeficiency 13. Subject has a clinically relevant active infection (eg. sepsis, pneumonia, and abscess) or has had a serious infection (resulting in hospitalization or parenteral antibiotic treatment) within 6 weeks prior to the first dose of rituximab.

14. Subject has an active neoplastic disease or history of neoplastic disease within 5 years of study entry (except for basal or squamous cell carcinoma of the skin or carcinoma in situ of the uterine cervix which has been definitely treated with standard of care approaches).

15. Subject was treated with plasma exchange or immunoabsorption within one month before inclusion, with immunosuppressive/chemotherapeutic medications including azathioprine, cyclophosphamide, cyclosporine, mycophenolate, etanercept, methotrexate within 6 months before inclusion, other immunosuppressive medications (including mitoxantrone, alemtuzumab, cladribine, pimecrolimus , IPP-201101) at any time; total lymphoid irradiation or hematopoietic stem cell transplantation at any time; any biological therapy within 12 months before inclusion.

16. Subject has received a live vaccination within 8 weeks prior to the baseline visit or intends to have live vaccination during the course of the study or within 7 weeks following the final dose of rituximab.

17. Subject has had prior treatment with rituximab in the 12 months before inclusion 18. History of hypersensitivity to Rituximab or to drugs of similar chemical classes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Inflammatory Neuropathy Cause and Treatment (INCAT) Disability Scale | 6 months
  The proportion of patients with CIDP not responsive to conventional immune therapies that improve after therapy with rituximab
Medical Research Council sum score | 6 months
  The proportion of patients with CIDP not responsive to conventional immune therapies that improve after therapy with rituximab
Inflammatory Rasch-built Overall Disability Scale (I-RODS) | 6 months
  The proportion of patients with CIDP not responsive to conventional immune therapies that improve after therapy with rituximab

SECONDARY OUTCOMES:
Inflammatory Neuropathy Cause and Treatment (INCAT) Disability Scale | 12 months
  Proportion of patients with CIDP not responsive to conventional immune therapies that improve after therapy with rituximab
Medical Research Council sum score | 12 months
  Proportion of patients with CIDP not responsive to conventional immune therapies that improve after therapy with rituximab
Inflammatory Rasch-built Overall Disability Scale (I-RODS) | 12 months
  Proportion of patients with CIDP not responsive to conventional immune therapies that improve after therapy with rituximab
Treatment discontinuation | 12 months
  Proportion of patients discontinuing treatment with rituximab due to side effects or voluntary withdrawal or developing these effects within 12 months following treatment
Duration of clinical improvement after therapy with rituximab | 24 months
Proportion of patients that improve 6 and 12 months after therapy with rituximab in subgroups defined according to the presence or absence of antibody reactivities | 6 and 12 months
Proportion of patients that improve 6 and 12 months after therapy with rituximab in subgroups defined according to the CIDP clinical form (typical or atypical) | 6 and 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Clinico Humanitas, Rozzano, Milano, Italy

REFERENCES:
- [Derived] Doneddu PE, Cocito D, Fazio R, Benedetti L, Peci E, Liberatore G, Falzone YM, Germano F, Gallia F, Giannotta C, Lleixa C, Bianchi E, Nobile-Orazio E. Prospective open-label trial with rituximab in patients with chronic inflammatory demyelinating polyradiculoneuropathy not responding to conventional immune therapies. J Neurol Neurosurg Psychiatry. 2024 Aug 16;95(9):838-844. doi: 10.1136/jnnp-2023-332844. PMID 38729746